CLINICAL TRIAL: NCT02030847
Title: Phase II Study of Redirected Autologous T Cells Engineered to Contain Anti-CD19 Attached to TCR and 4-1BB Signaling Domains in Patients With Chemotherapy Resistant or RefractoryAcute Lymphoblastic Leukemia
Brief Title: Study of Redirected Autologous T Cells Engineered to Contain Anti-CD19 Attached to TCR and 4-1BB Signaling Domains in Patients With Chemotherapy Resistant or Refractory Acute Lymphoblastic Leukemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UPCC 21413, 818626
Record Dates: First submitted 2014-01-07; First posted 2014-01-09 (Estimated); Results first posted 2019-05-24 (Actual); Last update posted 2023-06-22 (Actual); Status verified 2019-08

CONDITIONS: Patients With B Cell ALL, Relapsed or Refractory, With no Available Curative Treatment Options
MeSH Terms: conditions — Recurrence | interventions — CTL019 chimeric antigen receptor

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Arm1 (Experimental): phase II study to determine the efficacy and safety of a single infusion of autologous T cells expressing CD19 chimeric antigen receptors expressing tandem TCRζ and 4-1BB (TCRζ/4-1BB) co-stimulatory domains (referred to as "CART-19" cells) in adult patients with relapsed or refractory B-cell acute lymphoblastic leukemia.
  Interventions: Biological: CART-19

INTERVENTIONS:
Biological: CART-19 — CART-19 cells transduced with a lentiviral vector to express anti-CD19 scFv TCR:41BB administered by a single i.v. infusion of 1 to 5 x 10^8 transduced CAR T cells
Biological: CART-19 — As of June 2014, dose was reduced to a single dose of 1-5x10^7 CART-19 cells.
Biological: CART-19 — In the protocol amendment in November 2014, the dose remained 1-5 x 10^7 CART-19 cells, but was revised to be administered via split dosing: 10% on Day 1, 30% on Day 2, 60% on Day 3.
Biological: CART-19 — In the protocol amendment in May 2015, the dose was changed to 1-5 x 10^8 CART-19 cells administered via split dosing: 10% on Day 1 (1-5x10^7), 30% on Day 2 (3x10^7-1.5x10^8), 60% on Day 3 (6x10^7-3x10^8).

SUMMARY:
This is a single center, single arm, open-label phase II study to determine the efficacy and safety of a single infusion of autologous T cells expressing CD19 chimeric antigen receptors expressing tandem TCR and 4-1BB (TCR/4-1BB) co-stimulatory domains (referred to as CART-19 cells) in adult patients with relapsed or refractory B-cell acute lymphoblastic leukemia. Inclusion criteria are designed to include adult patients aged greater than 18 with B cell ALL, relapsed or refractory, with no available curative treatment options (such as autologous or allogeneic stem cell transplantation) who have limited prognosis (greater than 12 weeks survival expectancy) with currently available therapies. The study product is CART-19 cells transduced with a lentiviral vector to express anti-CD19 scFv TCR:41BB administered by a single i.v. infusion of 1 to 5 x 108 transduced CAR T cells.

ELIGIBILITY:
Inclusion Criteria

* Signed informed consent form must be obtained prior to any study procedure
* Relapsed or refractory B-cell ALL

  1. 1st or greater BM relapse OR
  2. Any marrow relapse after allogeneic HSCT and > 100 days from transplant OR
  3. For patients with refractory disease:

  i. < 60 years old that have not achieved a CR after > 2 or more chemotherapy regimens ii. >60 years old that have not achieved a CR after 1 prior chemotherapy regimen d. Patients with Ph+ ALL are eligible if they have failed tyrosine kinase inhibitor therapy
* Documentation of CD19 tumor expression in bone marrow or peripheral blood by flow cytometry within 3 months of screening.
* Adequate organ function defined as:

  1. Creatinine < 1.6 mg/dl
  2. ALT/AST < 3x upper limit of normal range
  3. Direct bilirubin <2.0 mg/dl
  4. Must have a minimum level of pulmonary reserve defined as ≤ Grade 1 dyspnea, pulse oxygen > 92% on room air, and DLCO > 40% (corrected for anemia if clinically appropriate)
  5. Left Ventricle Ejection Fraction (LVEF) ≥ 40% confirmed by ECHO/MUGA
* Bone marrow with ≥ 5% lymphoblasts
* Male or female age ≥ 18 years
* A ECOG Performance Status that is either 0 or 1
* No contraindications for leukapheresis.

Retreatment Inclusion Criteria

* Performance Status 0-1
* Adequate organ system function including:

  * Creatinine < 1.6 mg/dl
  * ALT/AST < 3x upper limit of normal
  * Total Bilirubin < 2.0 mg/dl
  * Must have a minimum level of pulmonary reserve defined as ≤ Grade 1 dyspnea, pulse oxygen > 92% on room air, and DLCO > 40% (corrected for anemia if clinically appropriate)
* Left Ventricular Ejection Fraction ≥ 40%
* No contraindications for leukapheresis (if required for retreatment)
* Gives voluntary informed consent for retreatment

Exclusion Criteria

* Isolated extramedullary disease relapse
* Active hepatitis B or active hepatitis C
* Class III/IV cardiovascular disability according to the New York Heart Association Classification
* HIV infection
* Active acute or chronic graft-versus-host disease (GVHD) or requirement of immunosuppressant medications for GVHD within 4 weeks of enrollment.
* Concurrent use of systemic steroids or chronic use of immunosuppressant medications. Recent or current use of inhaled steroids is not exclusionary. For additional details regarding use of steroid and immunosuppressant medications.
* Active CNS involvement by malignancy. Note: Patients with history of CNS disease that has been effectively treated will be eligible provided that treatment was >4 weeks before enrollment
* Pregnant or nursing (lactating) women, female study participants of reproductive potential must have a negative serum or urine pregnancy test within 48 hours before infusion
* Participation in a prior investigational study within 4 weeks prior to enrollment or longer if required by local regulation. Participation in non-therapeutic research studies is allowed.
* Patients with a known history or prior diagnosis of optic neuritis or other immunologic or inflammatory disease affecting the central nervous system.

Retreatment Exclusion Criteria

* Pregnant or lactating women.
* Active hepatitis B or hepatitis C
* Concurrent use of systemic steroids or chronic use of immunosuppressant medications. Recent or current use of inhaled steroids is not exclusionary. For additional details regarding use of steroid or immunosuppressant medications.
* HIV infection
* Patients with active CNS involvement with malignancy. Patients with prior CNS disease that has been effectively treated will be eligible providing treatment was >4 weeks before enrollment on the retreatment cohort.
* Class III/IV cardiovascular disability according to the New York Heart Association Classification
* Patients with a known history or prior diagnosis of optic neuritis or other immunologic or inflammatory disease affecting the central nervous system.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2014-02-27 (Actual); Primary Completion 2018-04-26 (Actual); Study Completion 2018-04-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Noelle Frey, MD, Principal Investigator — Abramson Cancer Center at Penn Medicine
Locations (1):
- Abramson Cancer Center of the University of Pennsylvania, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Derived] Frey NV, Shaw PA, Hexner EO, Pequignot E, Gill S, Luger SM, Mangan JK, Loren AW, Perl AE, Maude SL, Grupp SA, Shah NN, Gilmore J, Lacey SF, Melenhorst JJ, Levine BL, June CH, Porter DL. Optimizing Chimeric Antigen Receptor T-Cell Therapy for Adults With Acute Lymphoblastic Leukemia. J Clin Oncol. 2020 Feb 10;38(5):415-422. doi: 10.1200/JCO.19.01892. Epub 2019 Dec 9. PMID 31815579

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were identified through the clinical practices of the investigator or sub-investigators and through referrals from outside hospitals and physicians. No direct-to-patient advertising was performed.
Groups:
- Arm1: Phase II study to determine the efficacy & safety of a single infusion of autologous T cells expressing CD19 chimeric antigen receptors expressing tandem TCRζ and 4-1BB (TCRζ/4-1BB) co-stimulatory domains (referred to as "CART-19" cells) in adult patients with relapsed or refractory B-cell acute lymphoblastic leukemia.
  CART-19: CART-19 cells transduced with a lentiviral vector to express anti-CD19 scFv TCR:41BB administered by a single i.v. infusion of 1 to 5 x 10^8 transduced CAR T cells
  CART-19: As of June 2014, dose was reduced to a single dose of 1-5x10^7 CART-19 cells.
  CART-19: In the protocol amendment in November 2014, the dose remained 1-5 x 10^7 CART-19 cells, but was revised to be administered via split dosing: 10% on Day 1, 30% on Day 2, 60% on Day 3.
  CART-19: In the protocol amendment in May 2015, the dose was changed to 1-5 x 10^8 CART-19 cells administered via split dosing: 10% on Day 1 (1-5x10^7), 30% on Day 2 (3x10^7-1.5x10^8), 60% on Day 3 (6x10^7-3x10^8
Period: Overall Study
Arm/Group | Arm1
Started | 42
Completed | 5
Not Completed | 37
Not completed — Death | 10
Not completed — Disease Progression | 15
Not completed — New Cancer Therapy | 8
Not completed — Physician Decision | 3
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Population: Out of 42 enrolled, only 30 patients were infused with CART-19 product. 30 infused patients were considered for baseline analysis.
Arm/Group | Arm1
Number analyzed (Participants) | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.6 (16.34)
Age, Customized [Number; unit: participants]
  >=18 to <40 Years | 18
  >=40 to <65 Years | 10
  >=65 Years | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 20
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 28
  Unknown or Not Reported | 0
Race/Ethnicity, Customized [Number; unit: participants]
  Caucasian | 28
  Asian | 1
  Other | 1

OUTCOME MEASURES:

1. Primary Outcome: Overall Complete Remission Rate at Day 28 After CART-19 Therapy
Description: Overall Complete Remission Rate (ORR) which includes complete remission (CR) and CR with incomplete blood count recovery (CRi) at Day 28.
  Overall Complete Remission Rate = CR+ CRi
Time Frame: 28 Days
Population: Out of 42 enrolled, only 30 patients were infused with CART-19 product. 30 infused patients were considered for outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm1
Number analyzed (Participants) | 30
Participants
  Complete Remission (CR) | 8
  CR with incomplete blood count recovery (CRi) | 10
  No Response | 6
  Unknown | 6

2. Secondary Outcome: Best Overall Response
Description: For the secondary efficacy objectives for this study, the number of patients were computed with a best overall disease response of CR or CRi, where the best overall disease response is defined as the best disease response recorded from the start of the treatment until death, last follow up, relapse or start of new anticancer therapy, whichever comes first.
Time Frame: from the start of the treatment until death, last follow up, relapse or start of new anticancer therapy, whichever comes first, assessed up to 12 months
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Groups:
- Arm1: Phase II study to determine the efficacy & safety of a single infusion of autologous T cells expressing CD19 chimeric antigen receptors expressing tandem TCRζ and 4-1BB (TCRζ/4-1BB) co-stimulatory domains (referred to as "CART-19" cells) in adult patients with relapsed or refractory B-cell acute lymphoblastic leukemia.
  CART-19: CART-19 cells transduced with a lentiviral vector to express anti-CD19 scFv TCR:41BB administered by a single i.v. infusion of 1 to 5 x 10^8 transduced CAR T cells
  CART-19: As of June 2014, dose was reduced to a single dose of 1-5x10^7 CART-19 cells.
  CART-19: In the protocol amendment in November 2014, the dose remained 1-5 x 10^7 CART-19 cells, but was revised to be administered via split dosing: 10% on Day 1, 30% on Day 2, 60% on Day 3.
  CART-19: In the protocol amendment in May 2015, the dose was changed to 1-5 x 10^8 CART-19 cells administered via split dosing: 10% on Day 1 (1-5x10^7), 30% on Day 2 (3x10^7-1.5x10^8), 60% on Day 3 (6x10^7-3x10^8).
Arm/Group | Arm1
Number analyzed (Participants) | 30
Participants
  Complete Remission (CR) | 10
  CR with incomplete blood count recovery (CRi) | 1
  No Response | 8
  Unknown | 11

ADVERSE EVENTS:
Time Frame: 12 Months
Description: The remaining 12 participants that did not receive IP were not included in the AE Reporting, causing only 30 / 42 to be at risk".
Groups:
- Arm1: Phase II study to determine the efficacy & safety of a single infusion of autologous T cells expressing CD19 chimeric antigen receptors expressing tandem TCRζ & 4-1BB (TCRζ/4-1BB) co-stimulatory domains (referred to as "CART-19" cells) in adult patients with relapsed or refractory B-cell acute lymphoblastic leukemia.
  CART-19: CART-19 cells transduced with a lentiviral vector to express anti-CD19 scFv TCR:41BB administered by a single i.v. infusion of 1 to 5 x 10^8 transduced CAR T cells.
  CART-19: As of June 2014, dose was reduced to a single dose of 1-5x10^7 CART-19 cells.
  CART-19: In the protocol amendment in November 2014, the dose remained 1-5 x 10^7 CART-19 cells, but was revised to be administered via split dosing: 10% on Day 1, 30% on Day 2, 60% on Day 3.
  CART-19: In the protocol amendment in May 2015, the dose was changed to 1-5 x 10^8 CART-19 cells administered via split dosing: 10% on Day 1 (1-5x10^7), 30% on Day 2 (3x10^7-1.5x10^8), 60% on Day 3 (6x10^7-3x10^8).
Arm/Group | Arm1
All-Cause Mortality (participants affected / at risk) | 30/42
Serious Adverse Events (participants affected / at risk) | 30/30
Other Adverse Events (participants affected / at risk) | 30/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm1 (N=30)
Cytokine Release Syndrome (Immune system disorders) | 21
Sepsis (Infections and infestations) | 3
Pneumonia (Infections and infestations) | 2
Acidosis (Metabolism and nutrition disorders) | 1
Clostridium difficile infection (Infections and infestations) | 1
Constipation (Gastrointestinal disorders) | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 1
Haemorrhage intracranial (Nervous system disorders) | 1
Headache (Nervous system disorders) | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1
Influenza (Infections and infestations) | 1
Meningitis (Infections and infestations) | 1
Seizure (Nervous system disorders) | 1
Staphylococcal infection (Infections and infestations) | 1
Suicide attempt (Psychiatric disorders) | 1
Vision blurred (Eye disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm1 (N=30)
Anemia (Blood and lymphatic system disorders) | 16
Thrombocytopenia (Blood and lymphatic system disorders) | 4
Febrile Neutropenia (Blood and lymphatic system disorders) | 2
Neutropenia (Blood and lymphatic system disorders) | 2
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 1
Pulseless electrical activity (Cardiac disorders) | 1
Sinus Tachycarida (Cardiac disorders) | 1
Tachycardia (Cardiac disorders) | 1
Ear Pain (Ear and labyrinth disorders) | 1
Eye haemorrhage (Eye disorders) | 1
Papilloedema (Eye disorders) | 1
Vision blurred (Eye disorders) | 1
Vitreous haemorrhage (Eye disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 4
Constipation (Gastrointestinal disorders) | 2
Nausea (Gastrointestinal disorders) | 2
Stomatitis (Gastrointestinal disorders) | 2
Vomiting (Gastrointestinal disorders) | 2
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1
Pancreatitis (Gastrointestinal disorders) | 1
Tomgue ulceration (Gastrointestinal disorders) | 1
Fatigue (General disorders) | 5
Oedema peripheral (General disorders) | 5
Chills (General disorders) | 4
Pyrexia (General disorders) | 4
Generalised Oedema (General disorders) | 1
Influenza like illness (General disorders) | 1
Medical device site pain (General disorders) | 1
Cytokine release syndrome (Immune system disorders) | 28
Sepsis (Infections and infestations) | 3
Clostridium difficile colitis (Infections and infestations) | 2
Pneumonia (Infections and infestations) | 2
Bacterial infection (Infections and infestations) | 1
Clostridium difficile infection (Infections and infestations) | 1
Enterocolitis infections (Infections and infestations) | 1
Influenza (Infections and infestations) | 1
Meningitis (Infections and infestations) | 1
Oral candidiasis (Infections and infestations) | 1
Staphylococoal infection (Infections and infestations) | 1
Vira upper respiratory tract infection (Infections and infestations) | 1
Tendon injury (Injury, poisoning and procedural complications) | 1
Thermal burn (Injury, poisoning and procedural complications) | 1
Alanine aminotransferase increased (Investigations) | 17
Asprtate aminotransferase increased (Investigations) | 17
Platelet count decreased (Investigations) | 13
Neurphil count decreased (Investigations) | 11
Blood bilirubin increased (Investigations) | 10
White blood cell count decreased (Investigations) | 9
Blood alkaline phosphate increased (Investigations) | 8
Lymmphocyte count decreased (Investigations) | 7
Blood fibrinogen decreased (Investigations) | 5
Activated partial thromboplastin time prolonged (Investigations) | 3
Cd4 lymphocytes decreased (Investigations) | 3
Alanine aminotransferase (Investigations) | 1
Blood creatinine increased (Investigations) | 1
Ejection fraction decreased (Investigations) | 1
Hypocalcaemia (Metabolism and nutrition disorders) | 21
Hypophosphotaemia (Metabolism and nutrition disorders) | 17
Hyponatraemia (Metabolism and nutrition disorders) | 16
Hypokalemia (Metabolism and nutrition disorders) | 14
Hypoalbuminaemia (Metabolism and nutrition disorders) | 12
Hypomagnesaemia (Metabolism and nutrition disorders) | 10
Decreased appetite (Metabolism and nutrition disorders) | 4
Hyperglycaemia (Metabolism and nutrition disorders) | 4
Hypermagnesaemia (Metabolism and nutrition disorders) | 3
Hypernatraemia (Metabolism and nutrition disorders) | 3
Acidosis (Metabolism and nutrition disorders) | 2
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 2
Hypercalcaemia (Metabolism and nutrition disorders) | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 1
Tumor lysis syndrom (Metabolism and nutrition disorders) | 1
Muscular wekness (Musculoskeletal and connective tissue disorders) | 3
Myalgia (Musculoskeletal and connective tissue disorders) | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 1
Muscle haemorrhage (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1
Pain in Jaw (Musculoskeletal and connective tissue disorders) | 1
Headache (Nervous system disorders) | 4
Seizure (Nervous system disorders) | 3
Dizziness (Nervous system disorders) | 1
Dysgeusia (Nervous system disorders) | 1
Encephalopathy (Nervous system disorders) | 1
Intracranial Haemorrhage (Nervous system disorders) | 1
Neuroptahy peripheral (Nervous system disorders) | 1
Mental status changes (Psychiatric disorders) | 4
Insomnia (Psychiatric disorders) | 3
Confusional state (Psychiatric disorders) | 2
Agitation (Psychiatric disorders) | 1
Delirium (Psychiatric disorders) | 1
Hellucination (Psychiatric disorders) | 1
Acute kidney injury (Renal and urinary disorders) | 5
Urinary incontinence (Renal and urinary disorders) | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 4
Cough (Respiratory, thoracic and mediastinal disorders) | 2
Dsypnoea (Respiratory, thoracic and mediastinal disorders) | 2
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1
Laryngeal haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1
Laryngeal oedema (Respiratory, thoracic and mediastinal disorders) | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1
Rash (Skin and subcutaneous tissue disorders) | 2
Ecchymosis (Skin and subcutaneous tissue disorders) | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1
Night sweats (Skin and subcutaneous tissue disorders) | 1
Rash erythematous (Skin and subcutaneous tissue disorders) | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1
Hypertension (Vascular disorders) | 2
Embolism venous (Vascular disorders) | 1
Hypotension (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-04-14): https://cdn.clinicaltrials.gov/large-docs/47/NCT02030847/Prot_SAP_001.pdf